CLINICAL TRIAL: NCT07144046
Title: The Effect of Long-term Micropore Coverage on Cosmetic Outcomes After Mastectomy
Brief Title: Tape Application Protocol for Enhanced Scars
Acronym: TAPES
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Gustav Gede Nervil, Principal Investigator, Herlev Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TAPES
Record Dates: First submitted 2025-08-11; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Scar Improvement; Cosmetic Outcome
Keywords: Cosmetic Scar Evaluation; Long term wound dressing; Scar formation; Mastectomy; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Micropore Filters

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Micropore tape (Active Comparator): Micropore covering of the medial half of the scar
  Interventions: Other: Micropore covering of the medial half of the scar
- Control (No Intervention): Standart Practice

INTERVENTIONS:
Other: Micropore covering of the medial half of the scar — 3 months of micropore covering of the medial half of the scar
  Other Names: Micropore
  Arms: Micropore tape

SUMMARY:
What is the purpose of this study? The Investigators want to find out whether applying Micropore surgical tape to the medial half of the mastectomy scar for 3 months helps improve its appearance after 12 months, compared to no intervention.

Why is this study important? Scars can cause discomfort and affect how people feel about their bodies. The tape is thought to reduce stress on healing skin and possibly lead to a better-looking scar. But The Investigators need strong evidence to know whether it really helps.

How will the study be done?

This is a randomized, observer-blinded trial.

Women having mastectomy are randomly assigned to either receive the tape on half their scar or receive no tape.

A plastic surgeon and a breast surgeon-who do not know which side had tape-will evaluate wounds using photos after 3 and 12 months.

Patients will also rate their scars using a questionnaire (POSAS), giving their personal view on color, thickness, stiffness, and symptoms like itch or pain.

What else are The Investigators looking at?

The Investigators will examine whether the treated half of the scar looks better than the untreated half within the same woman-this helps control for individual skin differences.

The Investigators will also compare treated versus untreated areas across different women to see if there is a consistent benefit.

If the untaped half of scars looks different from control scars, this may suggest differences between the groups that affect results.

What will this study reveal? It will show whether using the tape improves cosmetic outcomes after mastectomy, and whether patients and clinicians agree on how scars heal. The findings may guide better post-surgery care to reduce scars and improve confidence and quality of life.

DETAILED DESCRIPTION:
Detailed Description This study is a randomized, observer-blinded, controlled trial investigating whether application of Micropore surgical tape to the medial half of the mastectomy scar for three months results in improved long-term scar appearance compared to no intervention.

Background and Rationale Scarring after mastectomy can negatively affect body image, comfort, and quality of life. Various post-surgical dressings have been proposed to improve scar cosmesis, including paper-based adhesive tapes such as Micropore. The proposed mechanism is that such tapes may provide mechanical support to the healing wound, reduce tension across the incision, and create a stable microenvironment, thereby minimizing scar widening, irregularity, and discoloration.

While tape therapy is widely used in clinical practice, the evidence for its effectiveness in mastectomy scars is limited, and there is no consensus on its benefit in this context. This trial seeks to address this knowledge gap using a blinded photographic evaluation and patient-reported outcome measures.

Study Design

Participants are randomized in a 1:1 ratio to either:

Intervention group: Application of Micropore tape to the medial half of the mastectomy scar for three months, starting approximately three weeks after surgery.

Control group: No application of Micropore tape; the scar remains uncovered after suture removal.

Block randomization in blocks of four will be used to maintain balanced group sizes over the course of enrollment. Randomization will be performed in REDCap, and allocation will occur after written informed consent is obtained.

Blinding Scar assessments will be conducted by two independent observers (a plastic surgeon and a breast surgeon) who are blinded to group allocation. Evaluations are based on standardized photographs taken at 3 and 12 months postoperatively. Medial and lateral halves of each scar will be assessed separately.

The lateral half of the scar in the intervention group is untreated and is expected to be comparable to the entire scar in the control group. Differences in lateral-half scores between groups will be examined to detect any systematic group imbalances.

Outcome Measures

Primary endpoint:

Difference in scar cosmesis at 12 months between intervention and control groups, based on the SCAR scale (observer-rated) and the Patient and Observer Scar Assessment Scale (POSAS, patient-reported component).

Secondary endpoints:

Within-subject difference between medial and lateral halves of the scar (intraindividual comparison).

Change in scores from 3 to 12 months for both observer and patient assessments.

Assessment of potential systematic differences between groups by comparing lateral halves across arms.

Concordance analysis between patient-reported scores (POSAS) and clinician-rated scores (SCAR) to evaluate agreement and identify systematic bias.

Follow-Up and Data Collection

At 3 months:

Standardized photographs

Patient questionnaire (POSAS)

Compliance assessment for the intervention group

At 12 months:

Standardized photographs

Patient questionnaire (POSAS)

Observer ratings (SCAR scale) of medial and lateral halves from photographs

Photographs are taken under standardized conditions: fixed camera distance (100 cm), controlled lighting, neutral background, and frontal plus 45° angled views.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing mastectomi without primary recontruction
* BMI between 18-5 and 35
* Age between 18 and 80

Exclusion Criteria:

* Known bandaid allergy
* In need of Mepilex Border OP after surgery
* Concurrent treatment with systemic steroid treatment or other immunosuppresants
* Post surgical haematoma that requires surgical intervention
* Known tendency to kelloid or hypertrophic scar formation

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
SCAR score after 1 year | 1 year
  Blinded observer score using The Scar Cosmesis Assessment and Rating (SCAR) scale to score surgical scar outcome from photos of the mastectomy incision at 12 months.

SECONDARY OUTCOMES:
POSAS Score at 12 months | 1 year
  Patient and Observer Reported Outcome using The Patient and Observer Scar Assessment Scale (POSAS) at 12 months after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Gustav Nervil, MD, PhD, Study Director

IPD SHARING:
Plan to Share IPD: Undecided
Danish Data legislation makes sharing of patient data that can be tracked back to the individual patient illigal.